CLINICAL TRIAL: NCT06665932
Title: Stereotactic Radiotherapy of Prostate Cancer With Reduction of Safety Margins
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONK-11-SBRT; 16/RVO-FNOs/2024 (Other Grant/Funding Number: University Hospital Ostrava)
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer (Adenocarcinoma)
Keywords: prostate cancer; Stereotactic Body Radiotherapy; acute toxicity; late toxicity
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Men with prostate cancer (Experimental)
  Interventions: Procedure: Stereotactic radiotherapy

INTERVENTIONS:
Procedure: Stereotactic radiotherapy — Stereotactic surgery is a minimally invasive form of surgical intervention that makes use of a three-dimensional coordinate system to locate small targets inside the body and to perform on them some action such as ablation, biopsy, lesion, injection, stimulation, implantation, radiosurgery, etc.

SUMMARY:
The study aims to reduce the PTV (Planning Target Volume) safety margins to 1-2 mm in stereotactic prostate radiotherapy for low- and medium-risk prostate cancers while maintaining a dose of 36.25 Gy in 5 fractions per day. By reducing the hems, the investigators expect a reduction of acute and late toxicity on the organs at risk, dominantly the urethra, bladder, penile bulb, and rectum, and an improvement in the quality of life.

DETAILED DESCRIPTION:
In this prospective study, a total of 100 patients will be treated over 2 years. Patients will be implanted with 4 contrast markers (fiducials) in the prostate - in the base, apex, and right and left lobes of the prostate. Subsequently, 3 planning examinations will be performed: 1. CT with a urinary catheter immediately after the implantation of fiducials (gold contrast markers), with a distance from implantation 2. planning CT and MR without a urinary catheter. The CTV (Clinical Target Volume) will be defined by the prostate, and the border on the PTV will be reduced from 3-5 mm to 1-2 mm isometrically to maximize the reduction of doses to the organs at risk (rectum, bladder, and urethra, penile bulb, testes), the organs at risk (OAR) will be marked in the radiation plan as OAR. Subsequently, the patients will be irradiated with a dose of 36.25 Gy in 5 fractions per day. Acute toxicity will be evaluated in the 1st and 3rd month after radiotherapy, and late toxicity after 4-6 months according to CTCAE criteria (Common Terminology Criteria for Adverse Events).

ELIGIBILITY:
Inclusion Criteria:

* histologically verified, localized prostate cancer without regional lymphadenopathy or distant metastases
* low or intermediate risk - favorable risk
* staging according to NCCN recommendations:
* low risk: no staging required
* intermediate risk- favorable risk: CT abdomen and pelvis
* PSA up to 15
* age over 18 years
* signed informed consent form
* suitable position of fiducials (to be determined by the physicist)

Exclusion Criteria:

* a histological type other than acinar adenocarcinoma
* the presence of local lymphadenopathy or distant metastases
* a dominant lesion in the periphery that is in contact with the capsule or grows through it
* PSA over 15
* unsatisfactory position of fiducials (to be determined by the physicist)
* previous treatment with radiotherapy to the pelvic area

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male patients with prostate cancer will be enrolled in the study.
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity incidence | 3 months from treatment
  Incidence of acute urological toxicity grade 2 and more according to the Common Terminology Criteria for Adverse Events (CTCAE) 4.03 scale
Acute toxicity of the lower gastrointestinal tract (GIT) | 3 months from treatment
  Incidence of acute toxicity of the lower GIT grade 2 and more according to the Common Terminology Criteria for Adverse Events (CTCAE) 4.03 scale

SECONDARY OUTCOMES:
5-year cumulative toxicity | 5 years
  5-year cumulative toxicity (urological and lower GIT) according to the CTCAE 4.03 scale
Quality of Life according to the EPIC-26 scale | 5 years from treatment
  Quality of Life will be assessed using the Expanded Prostate Cancer Index Composite (EPIC-26) scale
Quality of life (EQ-5D) | 5 years from treatment
  Quality of Life will be assessed using the EQ-5D tool

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
There is no plan to make individual participant data available to other researchers. The data may be provided upon request.

REFERENCES:
- [Background] Kishan AU, Ma TM, Lamb JM, Casado M, Wilhalme H, Low DA, Sheng K, Sharma S, Nickols NG, Pham J, Yang Y, Gao Y, Neylon J, Basehart V, Cao M, Steinberg ML. Magnetic Resonance Imaging-Guided vs Computed Tomography-Guided Stereotactic Body Radiotherapy for Prostate Cancer: The MIRAGE Randomized Clinical Trial. JAMA Oncol. 2023 Mar 1;9(3):365-373. doi: 10.1001/jamaoncol.2022.6558. PMID 36633877
- [Background] Dearnaley DP, Sydes MR, Graham JD, Aird EG, Bottomley D, Cowan RA, Huddart RA, Jose CC, Matthews JH, Millar J, Moore AR, Morgan RC, Russell JM, Scrase CD, Stephens RJ, Syndikus I, Parmar MK; RT01 collaborators. Escalated-dose versus standard-dose conformal radiotherapy in prostate cancer: first results from the MRC RT01 randomised controlled trial. Lancet Oncol. 2007 Jun;8(6):475-87. doi: 10.1016/S1470-2045(07)70143-2. PMID 17482880